CLINICAL TRIAL: NCT01084655
Title: An Open-label Phase 1/2 Study of TAK-700 in Combination With Docetaxel and Prednisone in Men With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of TAK-700 in Combination With Docetaxel and Prednisone in Men With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C21003
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone (Experimental): Orteronel (TAK-700) 200 milligram (mg), tablets, orally, twice daily (BID) starting from Day 1 along with docetaxel 75 milligram per square meter (mg/m^2), infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets , orally, twice daily from Day 8 up to Day 21 of each treatment cycle. Cycle 1 of Phase 1 consisted of a 28-day treatment period and subsequent cycles consisted of 21-day treatment periods.
  Interventions: Drug: TAK-700; Drug: Docetaxel; Drug: Prednisone
- Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone (Experimental): Orteronel (TAK-700) 400 mg, tablets, orally, twice daily starting from Day 1 along with docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets , orally, twice daily from Day 8 up to Day 21 of each treatment cycle. Cycle 1 of Phase 1 consisted of a 28-day treatment period and subsequent cycles consisted of 21-day treatment periods.
  Interventions: Drug: TAK-700; Drug: Docetaxel; Drug: Prednisone
- Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone (Experimental): Orteronel (TAK-700) 400 mg, tablets, orally, twice daily starting from Cycle 1 Day 15 along with docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets, orally, twice daily from Day 1 up to Day 21 of each 21-day treatment cycle until disease progression or end of treatment (EOT).
  Interventions: Drug: TAK-700; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: TAK-700 — TAK-700 with docetaxel and prednisone on a continuous schedule.
Drug: Docetaxel — TAK-700 with docetaxel and prednisone on a continuous schedule.
Drug: Prednisone — TAK-700 with docetaxel and prednisone on a continuous schedule.

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study of TAK-700 in combination with docetaxel and prednisone that will evaluate the safety and pharmacokinetics (PK) of the combination and will allow estimation of prostate-specific antigen (PSA) response in men with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria:

* Voluntary written consent
* Male patients 18 years or older
* Estimated life expectancy of 6 months or more
* Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma
* Radiograph-documented metastatic disease
* Progressive disease
* Prior surgical castration or concurrent use of an agent for medical castration
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Physical examination findings that are consistent with other study entry or exclusion criteria and identified but not excluded chronic conditions
* Even if surgically sterilized, patients must Practice effective barrier contraception during the entire study treatment period through 6 months after the last dose of study drug, OR Abstain from heterosexual intercourse
* Any use of opiates must be stable for at least 2 weeks prior to study entry
* Meet screening laboratory values as specified in protocol
* Suitable venous access

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Known hypersensitivity to TAK-700, docetaxel, prednisone or related compounds
* Received any of the following within 30 days prior to the first dose of TAK-700: prior therapy with any investigational compound; prior herbal product known to decrease PSA; OR radiation therapy for prostate cancer
* Received prior therapy with TAK-700, aminoglutethimide, ketoconazole or abiraterone (for Phase 1 only, patients previously treated with ketoconazole or abiraterone will be eligible if treatment with ketoconazole or abiraterone was discontinued at least 30 days prior to enrollment)
* Received antiandrogen therapy within 4 weeks for flutamide and 6 weeks for all others prior to first dose of study drug
* Received prior chemotherapy for prostate cancer
* Current spinal cord compression, bilateral hydronephrosis or neck outlet obstruction
* Symptoms that investigator deems related to prostate cancer
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Uncontrolled cardiovascular condition
* New York Heart Association Class (NYHA) Class III or IV
* Uncontrolled hypertension despite medical therapy
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Unwilling or unable to comply with protocol
* Major surgery or serious infection within 14 days of first dose of TAK-700
* Life-threatening illness unrelated to cancer
* Uncontrolled nausea, vomiting or diarrhea
* Known gastrointestinal disease or procedure that could interfere with oral absorption or tolerance of TAK-700

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-07; Primary Completion 2013-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Alaska Clinical Research Center, LLC, Anchorage, Alaska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in the United States from 22 July 2010 to 03 March 2016.
Pre-assignment Details: Male participants with a historical diagnosis of metastatic-castration resistant prostate cancer (mCRPC) were enrolled in this 2 part study to receive orteronel (TAK-700) along with docetaxel 75 milligram per square meter (mg/m^2) and prednisone 5 milligram (mg) twice daily (BID).
Groups:
- Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone: Orteronel (TAK-700) 200 mg, tablets, orally, twice daily starting from Day 1 along with docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets, orally, twice daily from Day 8 up to Day 21 of each treatment cycle. Cycle 1 of Phase 1 consisted of a 28-day treatment period and subsequent cycles consisted of 21-day treatment periods.
- Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone: Orteronel (TAK-700) 400 mg, tablets, orally, twice daily starting from Cycle 1 Day 15, then given continuously along with docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets, orally, twice daily from Day 1 up to Day 21 of each 21-day treatment cycle until disease progression or end of treatment (EOT).
Period: Overall Study
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Started | 6 | 8 | 24
Treated | 6 | 8 | 23
Completed | 0 | 2 | 5
Not Completed | 6 | 6 | 19
Not completed — Radiographic disease progression | 3 | 2 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 4
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Other | 0 | 3 | 2
Not completed — Symptomatic deterioration | 0 | 0 | 2
Not completed — Prostate-specificAntigen(PSA)progression | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone | Total
Number analyzed (Participants) | 6 | 8 | 23 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (9.20) | 65.3 (7.76) | 66.2 (9.21) | 66.6 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 8 | 23 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 6 | 7 | 22 | 35
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 6 | 21 | 32
  Black or African American | 1 | 2 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 23 | 37
Height [Mean (Standard Deviation); unit: centimeter] | 172.47 (8.150) | 179.39 (5.452) | 179.57 (6.684) | 178.38 (7.018)
Weight [Mean (Standard Deviation); unit: kilogram] | 89.08 (30.972) | 98.61 (20.296) | 101.83 (17.527) | 99.07 (20.557)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.525 (7.5049) | 30.589 (5.9713) | 31.599 (5.2488) | 31.044 (5.6762)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE) or Serious Adverse Events (SAE)
Time Frame: Baseline up to 30 days after last dose of study drug (Day of last dose for Phase 1: Cycle 84 Day 21; Phase 2: Cycle 48 Day 21)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Number; unit: participants
Groups:
- Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone: Orteronel (TAK-700) 200 mg, tablets, orally, twice daily starting from Day 1 along with docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets , orally, twice daily from Day 8 up to Day 21 of each treatment cycle. Cycle 1 of Phase 1 consisted of a 28-day treatment period and subsequent cycles consisted of 21-day treatment periods.
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 6 | 8 | 23
participants
  TEAE | 6 | 8 | 23
  SAE | 5 | 5 | 16

2. Primary Outcome: Number of Participants With TEAEs Related to Hematology and Serum Chemistry
Time Frame: as for outcome 1
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Number; unit: participants
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 6 | 8 | 23
participants
  Neutropenia | 3 | 4 | 8
  Anaemia | 2 | 0 | 6
  Leukopenia | 0 | 1 | 4
  Leukocytosis | 0 | 0 | 3
  Neutrophil count decreased | 1 | 2 | 4
  Blood bilirubin increased | 0 | 1 | 1
  Blood creatinine increased | 1 | 0 | 2
  White blood cell count decreased | 0 | 3 | 6
  Gamma-glutamyltransferase increased | 0 | 0 | 4
  Blood alkaline phosphatase increased | 0 | 0 | 3
  Alanine aminotransferase increased | 0 | 0 | 2
  Aspartate aminotransferase increased | 0 | 0 | 2
  Hyperglycaemia | 3 | 4 | 4
  Hypomagnesaemia | 1 | 2 | 3
  Hyponatraemia | 1 | 1 | 2
  Hypophosphataemia | 0 | 3 | 2
  Hyperkalaemia | 0 | 3 | 0

3. Primary Outcome: Number of Participants With TEAEs Related to Vital Signs
Time Frame: as for outcome 1
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Number; unit: participants
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 6 | 8 | 23
participants
  Hypertension | 3 | 2 | 1
  Hypotension | 1 | 0 | 1
  Accelerated hypertension | 0 | 0 | 1

4. Primary Outcome: Number of Participants With TEAEs Related to Electrocardiogram (ECG)
Time Frame: as for outcome 1
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Number; unit: participants
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 6 | 8 | 23
participants
  Overall | 1 | 0 | 1
  Angina pectoris | 1 | 0 | 1

5. Primary Outcome: Phase 2: Cmax: Maximum Observed Plasma Concentration for Docetaxel
Time Frame: Cycle 1 Day 1: pre-dose and at multiple time points (up to 24 hours) post-end of docetaxel infusion; Cycle 2 Day 1: pre-dose and at multiple time points (up to 8 hours) post-end of docetaxel infusion
Population: The pharmacokinetic (PK)-evaluable population included participants who had sufficient dosing data and plasma concentration-time data to permit calculation of at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg: Docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets, orally, twice daily from Day 1 up to Day 21 of Treatment Cycle 1.
- Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone: Orteronel (TAK-700) 400 mg, tablets, orally, twice daily starting from Day 1 along with docetaxel 75 mg/m^2, infusion, intravenously over 1 hour on Day 1 and prednisone 5 mg, tablets, orally, twice daily from Day 1 up to Day 21 of Treatment Cycle 2.
Arm/Group | Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg | Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 9 | 7
nanogram per milliliter (ng/mL) | 1330 (41.6) | 1600 (25.9)
Statistical Analysis 1: Comparison: Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg vs Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone; ANOVA with dose level as a fixed effect and participant as a random effect; Test type: Superiority or Other; Ratio of Geometric Least Square(LS)Means = 1.204, 90% CI 2-sided [0.870 to 1.666]

6. Primary Outcome: Phase 2: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Docetaxel
Time Frame: as for outcome 5
Population: The PK-evaluable population included participants who had sufficient dosing data and plasma concentration-time data to permit calculation of at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg | Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 9 | 7
nanogram*hour per milliliter (ng*hr/mL) | 1180 (43.7) | 1270 (25.0)
Statistical Analysis 1: Comparison: Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg vs Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone; ANOVA with dose level as a fixed effect and participant as a random effect; Test type: Superiority or Other; Ratio of Geometric LS Means = 1.074, 90% CI 2-sided [0.793 to 1.455]

7. Primary Outcome: Phase 2: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Docetaxel
Time Frame: as for outcome 5
Population: Data was not calculated since no participant was available for analysis.
Arm/Group | Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg | Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Phase 2: Terminal Phase Elimination Half-life (T1/2) for Docetaxel
Time Frame: as for outcome 5
Population: Data was not calculated since no participant was available for analysis.
Arm/Group | Phase 2 Cycle 1: Docetaxel 75 mg/m^2 + Prednisone 5 mg | Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Phase 2: Cmax, ss: Maximum Observed Plasma Concentration at Steady State for Orteronel
Time Frame: Cycle 1 Day 21: pre-dose and at multiple time points (up to 8 hours) post-dose for orteronel; Cycle 2 Day 1: pre-dose and at multiple time points (up to 8 hours) post-dose for orteronel
Population: PK set where Cmax,ss data was available. The PK-evaluable population included participants who had sufficient dosing data and plasma concentration-time data to permit calculation of at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Phase 2 Cycle 1: Orteronel 400 mg BID + Docetaxel + Prednisone: Orteronel 400 mg, tablets, orally, BID, on Day 21 of Treatment Cycle 1 along with docetaxel 75 mg/m^2, injection, intravenously on Day 1 and prednisone 5 mg, tablets, orally, BID from Day 1 up to Day 21 of Treatment Cycle 1.
Arm/Group | Phase 2 Cycle 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 7 | 5
ng/mL | 2660 (38.8) | 3000 (27.1)
Statistical Analysis 1: Comparison: Phase 2 Cycle 1: Orteronel 400 mg BID + Docetaxel + Prednisone vs Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone; ANOVA with dose level as a fixed effect and participant as a random effect; Test type: Superiority or Other; Ratio of Geometric LS Means = 1.066, 90% CI 2-sided [0.802 to 1.417]

10. Primary Outcome: Phase 2: AUC 0-tau: Area Under the Plasma Concentration Versus Time Curve Zero to the Time of the End of the Dosing Interval for Orteronel
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 2 Cycle 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 9 | 7
ng*hr/mL | 18000 (14.6) | 871 (44.9)
Statistical Analysis 1: Comparison: Phase 2 Cycle 1: Orteronel 400 mg BID + Docetaxel + Prednisone vs Phase 2 Cycle 2: Orteronel 400 mg BID + Docetaxel + Prednisone; ANOVA with dose level as a fixed effect and participant as a random effect; Test type: Superiority or Other; Ratio of Geometric LS Means = 1.068, 90% CI 2-sided [0.955 to 1.195]

11. Primary Outcome: Phase 2: Percentage of Participants With Prostate-specific Antigen (PSA) Response of 30 Percent (%), 50%, and 90%
Description: PSA response rates (PSA-30, PSA-50, and PSA-90) were defined as greater than or equal to (>=) 30%, 50%, and 90% reductions, respectively, from baseline in PSA concentration.
Time Frame: Cycle 4 Day 21
Population: The PSA-evaluable population included all participants with a baseline PSA evaluation and at least 1 PSA evaluation beyond Cycle 1, or participants with baseline PSA evaluation without a beyond-cycle-1 PSA evaluation due to PSA progression, disease progression, unacceptable adverse event (AE), or death.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 22
percentage of participants
  PSA-30 | 68 [52.3 to 81.3]
  PSA-50 | 59 [43.2 to 73.6]
  PSA-90 | 23 [11.5 to 38.1]

12. Primary Outcome: Phase 2: Best PSA Response
Description: Best PSA response was defined as the maximum PSA percent reduction from baseline at any time beyond Cycle 1.
Time Frame: Cycle 2 Day 1 up to Cycle 12 Day 21
Population: The PSA-evaluable population included all participants with a baseline PSA evaluation and at least 1 PSA evaluation beyond Cycle 1, or participants with baseline PSA evaluation without a beyond-cycle-1 PSA evaluation due to PSA progression, disease progression, unacceptable AE, or death.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 22
percent change | -61.72 (51.609) [11.5 to 38.1]

13. Secondary Outcome: Phase 2: Time to PSA Progression
Description: Time to PSA progression was defined as (date of PSA progression) - (date of first dose of drug) + 1, where PSA progression was defined as: For participants whose PSA concentrations never declined before the end of Cycle 4 of treatment: a) >=25% increase over the baseline level and an increase in absolute PSA concentration >=2 ng/mL; For participants who initially experienced a PSA decline: a) >=25% increase in PSA above the nadir concentration and an increase in absolute PSA concentration >=2 ng/mL.
Time Frame: Baseline until disease progression or death, whichever occurred first (up to approximately 25.4 months)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 23
days | 203 (51.609) [148.0 to 314.0]

14. Secondary Outcome: Phase 2: Time to Radiographic Disease Progression
Description: Time to Radiographic Disease Progression was defined as (date of Radiographic Disease progression) - (date of first dose of drug) + 1. Radiographic disease progression is defined as the presence of progressive disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1) criteria and/or bone scan progression determined according to second Prostate Cancer Clinical Trials Working Group (PCWG2) bone scan criteria.
Time Frame: Baseline until disease progression or death, whichever occurred first (up to approximately 25.4 months)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 23
days | 393 (51.609) [265.0 to NA] — Data was not estimable due to the low number of events in the arm.

15. Secondary Outcome: Phase 2: Percentage of Participants With Objective Measurable Disease Response
Description: Percentage of participants with objective measurable disease response based assessment of complete response (CR), partial response (PR), stable disease or PD according to RECIST (Version 1.1). A CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to less than (<)10 millimeter (mm). A PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of longest diameters of non-lymph node lesions and of the short diameter(s) or short axis of lymph nodes.
Time Frame: Baseline until disease progression or death, whichever occurred first (up to approximately 25.4 months)
Population: The RECIST-evaluable population was defined as all participants with measurable disease by RECIST (Version 1.1) at baseline, and with at least 1 postbaseline tumor response assessment (RECIST, Version 1.1).
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 10
percentage of participants
  Complete response | 0 (51.609) [44.8 to 88.4]
  Partial response | 70
  Stable Disease | 30
  Progressive Disease | 0

16. Secondary Outcome: Phase 2: Change From Baseline in Circulating Tumor Cells (CTCs)
Description: Baseline is defined as the last scheduled observed measurement prior to the first dose of drug.
Time Frame: Cycle 2 Day 1, Cycle 5 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1, Cycle 21 Day 1, End of treatment (approximately up to Cycle 48), Last assessment (30 days after last dose of study drug, approximately up to 1038 days)
Population: Safety analysis set where baseline and post-baseline assessments were available. The safety analysis set included all participants who were enrolled and received at least 1 dose of orteronel.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Number analyzed (Participants) | 21
milliliter (mL)
  Baseline (n=21) | 47.9 (108.85) [44.8 to 88.4]
  Change at Cycle 2 Day 1 (n=12) | -11.9 (24.57)
  Change at Cycle 5 Day 1 (n=16) | -39.0 (80.35)
  Change at Cycle 9 Day 1 (n=6) | -25.5 (35.07)
  Change at Cycle 13 Day 1 (n=7) | -11.3 (27.72)
  Change at Cycle 17 Day 1 (n=5) | -18.8 (31.93)
  Change at Cycle 21 Day 1 (n=1) | -5.0 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.
  Change at End of treatment (n=11) | -40.2 (66.43)
  Change at Last assessment (n=18) | -35.0 (76.30)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to Part 1: Cycle 29 Day 21; Part 2: Cycle 12 Day 21).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone
Serious Adverse Events (participants affected / at risk) | 5/6 | 5/8 | 16/23
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone (N=6) | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone (N=8) | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone (N=23)
Cellulitis (Infections and infestations) | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Orteronel 200 mg BID + Docetaxel + Prednisone (N=6) | Phase 1: Orteronel 400 mg BID + Docetaxel + Prednisone (N=8) | Phase 2: Orteronel 400 mg BID + Docetaxel + Prednisone (N=23)
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 8
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 3
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 11
Nausea (Gastrointestinal disorders) | 3 | 5 | 10
Constipation (Gastrointestinal disorders) | 3 | 2 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 5 | 8 | 17
Pyrexia (General disorders) | 1 | 2 | 4
Asthenia (General disorders) | 0 | 2 | 3
Oedema peripheral (General disorders) | 1 | 1 | 2
Chills (General disorders) | 1 | 1 | 1
Pain (General disorders) | 0 | 1 | 1
Peripheral swelling (General disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 2
Fungal skin infection (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Weight decreased (Investigations) | 2 | 3 | 4
White blood cell count decreased (Investigations) | 0 | 3 | 6
Neutrophil count decreased (Investigations) | 1 | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3
Blood creatinine increased (Investigations) | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 2
Ejection fraction decreased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 4 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 5
Dizziness (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 1 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 2 | 5
Anxiety (Psychiatric disorders) | 2 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 5
Dysuria (Renal and urinary disorders) | 0 | 0 | 4
Haematuria (Renal and urinary disorders) | 0 | 2 | 2
Nocturia (Renal and urinary disorders) | 1 | 2 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 6 | 14
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 3 | 2 | 2
Flushing (Vascular disorders) | 0 | 2 | 2
Hot flush (Vascular disorders) | 0 | 1 | 3
Hypotension (Vascular disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.